CLINICAL TRIAL: NCT05942326
Title: Sleep GOALS (Goal-focused Online Access to Lifestyle Support), an Internet Assisted Diet, Physical Activity, and Sleep Weight Loss Intervention for Postpartum Women
Brief Title: Sleep Goal-focused Online Access to Lifestyle Support
Acronym: SGOALS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Marquis Hawkins, Assistant Professor, University of Pittsburgh
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: STUDY23020169; K01HL161439 (NIH)
Record Dates: First submitted 2023-05-23; First posted 2023-07-12 (Actual); Last update posted 2025-04-11 (Actual); Status verified 2025-04

CONDITIONS: Weight Loss; Weight, Body
MeSH Terms: conditions — Weight Loss; Body Weight | interventions — Educational Status

STUDY DESIGN:
Intervention Model Description: 16-week pilot study will use a single-blind, parallel-arm randomized controlled trial design. Participants will be randomized at a 1:1 ratio to Sleep GOALS intervention (n=20) or an education control group (n=20)
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Sleep GOALS (Experimental): Weekly 15-to-20 minute educational video each, a commercial activity tracker (e.g., Fitbit) to monitor sleep and physical activity, wireless scale to monitor weight, and a lifestyle coach who will provide personalized support.
  Interventions: Behavioral: Sleep GOALS
- Education (Active Comparator): Brochures that provide tips for improving sleep health, diet, and physical activity
  Interventions: Behavioral: Education

INTERVENTIONS:
Behavioral: Sleep GOALS — Web-based interventions
  Arms: Sleep GOALS
Behavioral: Education — Brochures from the American Academy of Sleep Medicine (e.g., sleep hygiene, sleep in women) and SNAP education connection (e.g., family-friendly activities, meal planning)
  Arms: Education

SUMMARY:
The overall goal of the study is to develop a novel weight loss intervention for postpartum people by providing strategies to improve sleep, diet, and physical activity behaviors. In this study, we will recruitment and enroll 40 postpartum people and randomize them to receive the Sleep GOALS intervention or education control to evaluate the intervention's feasibility, acceptability, and preliminary efficacy.

ELIGIBILITY:
Inclusion Criteria:

* Stated willingness to comply with all study procedures and availability for the duration of the study,
* Primiparous, singleton pregnancy,
* Between 3+1 and 6+1 months postpartum,
* Has a body mass index >25 kg/m2,
* Physically inactive, defined as self-reporting <150 minutes/week of moderate-to-vigorous intensity physical activity,
* Endorse >1 indicator of poor sleep health based on the RU_SATED questionnaire, and
* Has smartphone and home Internet access

Exclusion Criteria:

* current use of medications that affect weight,
* currently pregnant or plan to become pregnant during the study period (18 weeks), and
* participating in another weight loss intervention.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2023-09-21 (Actual); Primary Completion 2025-01-22 (Actual); Study Completion 2025-01-22 (Actual)

PRIMARY OUTCOMES:
Recruitment/Enrollment - Number of the total sample | Baseline
  The number of participants enrolled in 12 months
Recruitment/Enrollment - Proportion of ethnic minority | Baseline
  The proportion of ethnic minority
Retention rates | Post-intervention at week 17
  1-Attrition rates, % with complete post-intervention data collection
Engagement - Number of modules completed | Week 1 to 16
  The number of modules completed within 16 weeks
Engagement - Number of self-monitoring of diet, sleep and physical activity weekly | Week 1 to 16
  The number of weeks in which self-monitoring of diet, sleep, and physical activity is performed at least once a week
Engagement - Number of weekly weigh-ins | Week 1 to 16
  The number of weeks in which weigh-in is performed at least once a week
Engagement - Total time logged in | Week 1 to 16
  Total time logged in during the 16-week intervention
Acceptability - Proportion of agreeing | Week 1 to Post-intervention at week 17
  Participant ratings on the intervention delivery; behavior change curricula; action plan; intervention platform.
  The questionnaire asks participants to provide answers on a 5-point scale (1=don't agree at all to 5=totally agree) to 39 items about the intervention delivery (e.g., logical, understandable), curricula (e.g., was it logical, relevant, instructive), action plans (e.g., useful, easy to follow), and intervention platform (e.g., user friendly).

SECONDARY OUTCOMES:
Weight change | Baseline and Post-intervention at week 17
  Baseline and post-intervention differences in weight. Weight will be measured with a digital scale, with the participant wearing light clothing and no shoes at baseline and post-intervention.
Postpartum weight retention | Post-intervention at week 17
  Pre-pregnancy and post-intervention differences in weight. Participants will self-report pre-pregnancy weight, and post-intervention weight will be measured with a digital scale, with the participant wearing light clothing and no shoes. The power-to-weight ratio (PWR) will be estimated as the difference in measured weight at post-intervention and self-reported pre-pregnancy weight.

CONTACTS AND LOCATIONS:
Overall Officials: Marquis Hawkins, PhD, Principal Investigator — University of Pittsburgh
Locations (1):
- University of Pittsburgh, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in the article after deidentification (text, tables, figures, and appendices)
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: Data will be made available after primary outcome manuscripts are published. Data will remain available in de-identified format with no end date specified.
Access Criteria: Data will be shared with investigators whose proposed use of the data has been approved by an independent review committee identified for this purpose. Researchers requesting use of data must submit their request in writing to the MPIs, including the purpose for which they are requesting use of the data. These requests will be reviewed by the Investigators and will require engaging in a Data Use Agreement (DUA), in cooperation with the University of Pittsburgh. Data will be shared to achieve aims in the approved proposal. We plan to use the Open Science generalist platform to share data, as requested. As the study is completed, we will share data using the NIDA data share website.

REFERENCES:
- [Derived] Hawkins MS, Davis EM, Abebe KZ, McTigue KM, Kim N, Goswami M, Buysse DJ, Chang JC, Levine MD. An internet-assisted sleep, dietary, and physical activity intervention to support weight-loss among postpartum people (Sleep GOALS): protocol for a pilot randomized controlled trial. Pilot Feasibility Stud. 2025 Nov 13;11(1):140. doi: 10.1186/s40814-025-01733-2. PMID 41233902